CLINICAL TRIAL: NCT00061763
Title: Phase II Study of Safety & Efficacy of Deferasirox Given for 1 Year in Patients With Chronic Anemias and Transfusional Hemosiderosis Unable to be Treated With Deferoxamine
Brief Title: Study of Deferasirox in Iron Overload From Beta-thalassemia Unable to be Treated With Deferoxamine or Chronic Anemias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A0108
Record Dates: First submitted 2003-06-03; First posted 2003-06-04 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Beta-thalassemia; Myelodysplastic Syndromes; Fanconi Syndrome; Anemia, Diamond-Blackfan; Anemia, Aplastic
Keywords: beta-thalassemia; iron overload; deferoxamine; Myelodysplastic Syndromes; Fanconi Syndrome; Anemia, Diamond-Blackfan; Anemia, Aplastic
MeSH Terms: conditions — beta-Thalassemia; Myelodysplastic Syndromes; Fanconi Syndrome; Anemia, Diamond-Blackfan; Anemia, Aplastic; Iron Overload | interventions — Deferasirox

INTERVENTIONS:
Drug: Deferasirox

SUMMARY:
The purpose of this study is to determine the effects of the oral iron chelator Deferasirox on liver iron content after one year of treatment in patients with iron overload from repeated blood transfusions. Beta-thalassemia patients unable to be treated with deferoxamine or patients with rare chronic anemias such as Myelodysplastic Syndrome, Fanconi's Syndrome, Blackfan-Diamond Syndrome, and Pure Red Blood Cell Anemia are eligible for this study. Liver iron content will be measured by liver biopsy at the beginning of the study and after one year of treatment. However, those patients living in the San Francisco/Oakland area may have a SQUID in place of the liver biopsy if the biopsy is not medically possible for them. The SQUID is a non-invasive magnetic means to measure liver iron content.

ELIGIBILITY:
Inclusion Criteria:

* Beta-thalassemia patients with documented non-compliance to deferoxamine, defined as taking less than 50% of prescribed doses in year prior to study, and having a liver iron content at least 14 mg iron/gm dry weight liver tissue
* Beta-thalassemia patients unable to take deferoxamine because of documented side effects or contra-indication, or documented poor response despite proper compliance, with liver iron content at least 2 mg iron/gm dry weight liver tissue
* Patients with chronic anemias with a liver iron content at least 2 mg/gm dry weight liver tissue.
* Beta-thalassemia or other chronic anemia patients having previously taken deferiprone, provided that they stop the deferiprone at least 28 days before the study and have a liver iron content at least 2 mg/gm dry weight liver tissue.
* All patients: Regular transfusions indicated by a requirement of at least 8 blood transfusions per year.
* Life expectancy of at least one year.

Exclusion Criteria:

* Beta-thalassemia able to be treated with deferoxamine, Sickle Cell Disease or non-transfusional iron overload
* Elevated liver enzymes in the year preceding enrollment
* Active Hepatitis B or Hepatitis C
* HIV seropositivity
* Elevated serum creatinine or significant proteinuria
* History of nephrotic syndrome
* Uncontrolled systemic hypertension
* Fever and other signs/symptoms of infection within 10 days prior to start of the study.
* Presence of clinically relevant cataract or previous history of clinically relevant ocular toxicity related to iron chelation.
* Second or third degree AV block, clinically relevant Q-T interval prolongation, or patients requiring digoxin or other drugs that prolong the Q-T interval.
* Diseases (cardiovascular, renal, hepatic, etc.) that would prevent the patient from undergoing any of the treatment options.
* Psychiatric or additive disorders that would prevent the patient from giving informed consent.
* History of drug or alcohol abuse within the 12 months prior to the study.
* Pregnant or breast feeding patients.
* Patients treated with systemic investigational drugs within 4 weeks or topical investigational drugs within 7 days before the start of teh study.
* Any surgical or medical condition that might significantly alter the absorption, distribution, metabolism or excretion of any drug, such as gastrointestinal disease or major surgery, renal disease, difficulty voiding or urinary obstruction, or impaired pancreatic function.
* Non-compliant or unreliable patients
* Patients unable to undergo any study procedures such as the hearing or eye tests, or the liver echocardiography.
* Patients that would need a dose of Deferasirox less than 125 mg per day.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2003-05; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of treatment on the liver iron content(LIC)

SECONDARY OUTCOMES:
Evaluate tolerability profile
Estimate the absolute and relative change of LIC and total body iron excretion (TBIE) rate
Evaluate the relationship between LIC and potential surrogate markers
Evaluate the relationship between PD and safety variables

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - Children's Hospital Oakland, Oakland, California
  - Stanford Hospital, Stanford, California
  - Northwest Medical Specialists, Arlington Heights, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Weill Medical College of Cornell University, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania